CLINICAL TRIAL: NCT00841100
Title: Kuvan Therapy in Phenylketonuria (PKU): The Effect of Blood Phenylalanine Concentration on Kuvan Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20080675
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Phenylketonuria
Keywords: PKU; Kuvan; BH4; tetrahydrobiopterin
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Acute 24 Hour Component (Experimental): Participants will receive one dose of Kuvan 20 mg/kg on Day 1 and assessed for Acute 24 hour Kuvan response.
  Interventions: Drug: Kuvan
- Phase 1 Group (Experimental): After completion of acute 24 hour component, participants can enroll in Phase 1 and will receive Kuvan 20 mg/kg by mouth once daily for 28 consecutive days
  Interventions: Drug: Kuvan
- Phase 2 Group (Experimental): Participants in Phase 1 that was not responsive will continue on to the Phase 2 of the study. Positive response is defined as a decrease of blood phenylalanine of 30% or greater from baseline taken from morning blood serum. The Phase 2 component of the study will be a 2 week period of dietary restriction.
  Interventions: Other: Diet
- Phase 3 Group (Experimental): Participants in Phase 2 that achieves a fasting blood phenylalanine of less than 600 umol/l after 2 week dietary restriction will be retreated with Kuvan 20 mg/kg by mouth once daily for a period of 28 consecutive days.
  Interventions: Drug: Kuvan

INTERVENTIONS:
Drug: Kuvan — 20mg/kg by mouth once daily
  Other Names: sapropterin dihydrochloride, Tetrahydrobiopterin (BH4)
  Arms: Acute 24 Hour Component; Phase 1 Group; Phase 3 Group
Other: Diet — Phenylalanine-restricted diet (4-10 mg/kg/day phenylalanine) using the prescribed phenylalanine-free medical formula and low protein foods tested with the patients for taste and acceptance to lower blood phenylalanine levels below 600 umol/l.
  Arms: Phase 2 Group

SUMMARY:
The investigators will investigate the effect of blood phenylalanine on Kuvan responsiveness in the same patients with PKU when their blood phenylalanine concentrations are altered by diet.

Lowering blood phenylalanine concentrations in Kuvan non-responsive patients with PKU will increase the frequency of Kuvan responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a diagnosis of phenylketonuria
* patients who are over the age of 4 years,
* patients with a fasting blood phenylalanine ≥600µmol/l

Exclusion Criteria:

* female patients who are pregnant or attempting to become pregnant
* children under four years of age
* Concurrent disease of condition that would interfere with study participation or safety such as history of neurological compromise or major medical, psychiatric or learning disorder unrelated to PKU
* Any condition that, in the view of the Investigators, places subject at high risk of poor treatment compliance or of not completing the study
* Use of L-Dopa, methotrexate, or other drugs that may inhibit folate metabolism

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2011-07-19 (Actual); Study Completion 2011-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Elsas, MD, Principal Investigator — University of Miami
Locations (1):
- Department of Biochemistry & Molecular Biology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton BK, Grange DK, Milanowski A, Vockley G, Feillet F, Crombez EA, Abadie V, Harding CO, Cederbaum S, Dobbelaere D, Smith A, Dorenbaum A. The response of patients with phenylketonuria and elevated serum phenylalanine to treatment with oral sapropterin dihydrochloride (6R-tetrahydrobiopterin): a phase II, multicentre, open-label, screening study. J Inherit Metab Dis. 2007 Oct;30(5):700-7. doi: 10.1007/s10545-007-0605-z. Epub 2007 Sep 12. PMID 17846916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants enrolled in the acute phase were eligible to continue onto the Phase 1 component of the trial. Only the participants who were non-responsive on the Phase 1 component of the study continued on to Phase 2. Only Phase 2 participants who achieved a fasting blood phenylalanine of less than 600 umol/l can continue to Phase 3.
Groups:
- All Participants: All participants were enrolled into the four arms of the study. The 24-hour component consisted of participants received one dose of Kuvan 20 mg/kg on Day 1 and assessed for Acute 24 hour Kuvan response. The Phase 1 arm consisted of participants who after completion of the acute 24-hour component, enrolled and received Kuvan 20 mg/kg by mouth once daily for 28 consecutive days. The Phase 2 arm consisted of participants in Phase 1 that were not responsive and continued on to Phase 2 of the study. Positive response is defined as a decrease of blood phenylalanine of 30% or greater from baseline taken from morning blood serum. The Phase 2 component of the study will be a 2 week period of dietary restriction.
  The Phase 3 arm of the study consisted of participants in Phase 2 that achieved a fasting blood phenylalanine of less than 600 umol/l after 2-week dietary restriction will be retreated with Kuvan 20 mg/kg by mouth once daily for a period of 28 consecutive days.
Period: Acute Component (24 Hours)
Arm/Group | All Participants
Started | 21
Completed | 21
Not Completed | 0
Period: Phase 1 (28 Days)
Arm/Group | All Participants
Started | 18 (3 participants from the acute phase elected not to continue to the Phase 1 component of the study.)
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Participant non-compliance | 2
Period: Phase 2 (2 Weeks)
Arm/Group | All Participants
Started | 5 (Participants who were non-responsive on the Phase 1 component of the study continued on to Phase 2.)
Completed | 5
Not Completed | 0
Period: Phase 3 (28 Days)
Arm/Group | All Participants
Started | 4 (Participants who achieved a fasting blood phenylalanine of <600 umol/l can continue to Phase 3.)
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that was enrolled in the study
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Blood Phenylalanine
Description: Percent change in phenylalanine in (uM) on Kuvan Response evaluated via fasting morning blood serum. A decrease of 30% or greater indicates positive response on Kuvan.
Time Frame: Baseline to Day 1 of the Acute Phase, Baseline to Day 28 of Phase 1, Baseline to Day 28 of Phase 3
Population: 3 participants from the acute phase elected not to continue to the Phase 1 component of the study. Participants who were non-responsive on the Phase 1 component of the study continued on to Phase 2. Participants who achieved a fasting blood phenylalanine of <600 umol/l can in Phase 2, continued to Phase 3.
Measure: Mean (Standard Deviation); unit: Percent change in blood phenylalanine
Groups:
- Ove.Erall Participants: All participants enrolled in the study.
Arm/Group | Ove.Erall Participants
Number analyzed (Participants) | 21
Percent change in blood phenylalanine
  Baseline to Day 1 of the Acute phase | -13.71 (21.62)
  Baseline to Day 28 of Phase 1: number analyzed (Participants) | 15
  Baseline to Day 28 of Phase 1 | -8.13 (31.84)
  Baseline to Day 28 of Phase 3: number analyzed (Participants) | 4
  Baseline to Day 28 of Phase 3 | 48.75 (61.87)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=21)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes